CLINICAL TRIAL: NCT06359054
Title: The Role of 68GA DOTATATE PET/CT In Breast Cancer Imaging; a Prospective Study Compared With 18F FDG PET/CT
Brief Title: The Role of 68GA DOTATATE PET/CT In Breast Cancer Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CelalBayarNRG
Record Dates: First submitted 2023-11-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breast Cancer Patient (Experimental)
  Interventions: Diagnostic Test: 18F FDG PET/CT; Diagnostic Test: 68Ga DOTATATE PET/CT

INTERVENTIONS:
Diagnostic Test: 18F FDG PET/CT — 18F-FDG PET/CT Imaging: Preparation: Participants will be instructed to fast for at least 6 hours before the procedure to ensure low insulin levels and high FDG uptake by cancer cells.
  Radiopharmaceutical Administration: Each participant will receive an intravenous injection of 18F-FDG, dosed at approximately 5.2 MBq/kg (0.14 mCi/kg) of body weight.
  Imaging Protocol: After the injection, participants will rest in a quiet and dimly lit room for approximately 60 minutes to allow for optimal distribution and uptake of 18F-FDG by the tissues. Subsequently, they will be positioned on the PET/CT scanner bed, and imaging will be performed from the vertex to the proximal thighs. The scan will include a low-dose CT for attenuation correction followed by PET imaging, with the acquisition time adjusted based on the specific protocol (typically 2-3 minutes per bed position).
Diagnostic Test: 68Ga DOTATATE PET/CT — 68Ga-DOTATATE PET/CT Imaging: Preparation: No specific fasting is required for 68Ga-DOTATATE PET/CT. However, participants may be advised to hydrate well before the procedure.
  Radiopharmaceutical Administration: Participants will receive an intravenous injection of 68Ga-DOTATATE, dosed at approximately 2.2 MBq/kg (0.06 mCi/kg) of body weight.
  Imaging Protocol: Similar to the 18F-FDG protocol, after receiving 68Ga-DOTATATE, participants will wait for about 60 minutes to allow for sufficient uptake of the tracer. They will then undergo PET/CT scanning in a supine position, covering the same body regions as the FDG scan. A low-dose CT scan will be conducted first for attenuation correction, followed by the PET scan, with acquisition parameters tailored to the optimal detection of somatostatin receptor expression.

SUMMARY:
Currently, F-18 FDG PET/CT is routinely used for breast cancer staging and treatment response assessment. Most breast cancers express Estrogen Receptor (ER) and Progesterone Receptor (PR) and this subtype shows lower activity on FDG imaging. 68Ga DOTATATE PET/CT is an effective imaging option for somatostatin receptor (SSTR) positive neuroendocrine tumors. There are case reports showing 68Ga DOTATATE uptake in non-Hodgkin lymphoma, meningioma, breast cancer, thyroid adenoma and papillary carcinoma. There are also histochemical studies showing that SSTR is a potential radiopharmaceutical target for ER+/PR+ breast cancer . Its hypothesized that 68Ga DOTATATE PET/CT may be superior to 18F FDG PET/CT primarily in hormone receptor (HR) positive breast cancer. In this study, its aimed to compare the uptake pattern of breast cancer lesions and HR status with 68Ga DOTATATE and 18F FDG uptake in lesions.

DETAILED DESCRIPTION:
This study is designed to explore and compare the uptake patterns of breast cancer lesions using two distinct PET/CT imaging modalities: 18F-FDG and 68Ga-DOTATATE. The primary goal is to assess the diagnostic and prognostic value of these imaging techniques in the context of breast cancer, with a particular focus on their ability to inform treatment strategies based on the biological characteristics and stage of the disease.

Breast cancer remains the most prevalent cancer among women globally, as highlighted by GLOBOCAN 2020 data. The disease's treatment involves a multifaceted approach, including surgery, chemotherapy, radiotherapy, targeted therapies, and endocrine therapy. The effectiveness of these treatments is significantly influenced by the tumor's biological attributes and its progression stage. In this light, the accurate pre-treatment staging of breast cancer is paramount, with 18F-FDG PET/CT playing an increasingly crucial role due to its high accuracy in detecting extra-axillary lymph node metastases and distant metastatic disease.

Somatostatin analogs, particularly 68Ga-DOTA-TATE, have emerged as potent tools for imaging and treating SSTR-positive neuroendocrine tumors, leveraging the high affinity of DOTA-TATE for SSTR2. This study extends the application of 68Ga-DOTATATE PET/CT to breast cancer, motivated by findings that SSTR2 is the most prevalent somatostatin receptor subtype in breast tumors. The differential expression of SSTR2, influenced by tumor differentiation and hormonal status, underlines the potential of 68Ga-DOTATATE PET/CT in providing additional insights into tumor biology.

The study will systematically compare the uptake of 18F-FDG and 68Ga-DOTATATE in breast cancer lesions, correlating these findings with histopathological subtypes and hormone receptor (ER and PR) as well as HER2 status. By doing so, it aims to elucidate the relevance of SSTR2 expression in the heterogeneity of breast cancer and its implications for targeting somatostatin receptors in diagnosis and therapy.

This research is expected to contribute significantly to the field of nuclear medicine and oncology by:

Providing comparative data on the diagnostic accuracy and prognostic value of 18F-FDG PET/CT and 68Ga-DOTATATE PET/CT in breast cancer staging.

Evaluating the expression of SSTR subtypes in breast cancer and their correlation with tumor histopathology and receptor status.

Assessing the potential of 68Ga-DOTATATE PET/CT as a complementary tool for the personalized management of breast cancer, particularly in cases with somatostatin receptor expression.

This study is guided by the latest advancements in molecular imaging and aims to refine breast cancer treatment protocols, offering a more tailored and effective approach to patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 90 years old
* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* Pathologically proven breast cancer by biopsy
* Patients must be able to understand the meaning of the study and sign the appropriate Ethical Committee approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Any medical or psychiatric condition that compromises the subject´s ability to participate in the study
* Any other significant disease including liver or renal disease
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Comparative Diagnostic Accuracy of 68Ga DOTATATE and 18F FDG PET/CT | The diagnostic accuracy will be assessed immediately following the completion of both PET/CT scans, with each participant undergoing both scans within a one-week interval. The analysis of images and interpretation of results will occur after all particip
  The primary outcome of this study is to assess and compare the diagnostic accuracy of 18F-FDG PET/CT and 68Ga-DOTATATE PET/CT in detecting primary and metastatic breast cancer lesions. This will be evaluated through the identification of lesion uptake patterns, quantified by the maximum standardized uptake value (SUVmax), and the presence of extra-axillary lymph node and distant metastases as indicated by each imaging modality.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Manisa Celal Bayar University Faculty of Medicine, General Surgery Department, Manisa
  - Manisa Celal Bayar University Faculty of Medicine, Nuclear Medicine Department, Manisa

REFERENCES:
- [Background] Guirguis MS, Adrada BE, Surasi DS, Dryden MJ. 68Ga-DOTATATE Uptake in Primary Breast Cancer. Clin Nucl Med. 2021 Mar 1;46(3):248-249. doi: 10.1097/RLU.0000000000003421. PMID 33234932